CLINICAL TRIAL: NCT00082797
Title: A Phase II Study Of Systemic High-Dose Methotrexate For The Treatment Of Glioblastoma Multiforme In Newly Diagnosed Patients With Measurable Disease
Brief Title: High-Dose Methotrexate and Leucovorin in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000360834; E1F02
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Leucovorin; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: leucovorin calcium
Drug: methotrexate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate, work in different ways to stop tumor cells from dividing so they stop growing or die. Leucovorin may decrease side effects caused by high-dose methotrexate.

PURPOSE: This phase II trial is studying how well giving high-dose methotrexate together with leucovorin works in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response in patients with newly diagnosed glioblastoma multiforme treated with high-dose methotrexate and leucovorin calcium.

Secondary

* Determine the acute toxicity of this regimen in these patients.
* Determine the duration of survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive high-dose methotrexate IV over 4 hours on day 1 and oral or IV leucovorin calcium every 6 hours beginning on day 2 and continuing until blood methotrexate levels are acceptable. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients then receive standard radiotherapy with or without chemotherapy. Patients with disease progression proceed to standard radiotherapy with or without chemotherapy upon stopping methotrexate therapy.

Patients are followed at 30 days and then every 2 months for up to 2 years.

PROJECTED ACCRUAL: A total of 19-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme (GBM)

  * Supratentorial grade IV disease
* Measurable and contrast-enhancing disease ≥ 1 cm by CT scan or MRI
* No radiographic evidence of ascites or pleural effusion

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGOT ≤ 4.0 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine ≤ 2.0 mg/dL
* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* No uncontrolled hypertension
* No unstable angina
* No symptomatic congestive heart failure
* No uncontrolled cardiac arrhythmia
* No myocardial infarction within the past 6 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to achieve hydration
* No diabetes insipidus
* No known hypersensitivity to methotrexate or leucovorin calcium
* No concurrent serious infection or medical illness that would preclude study participation
* No other malignancy within the past 2 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for GBM
* No prior administration of any of the following biologic agents for GBM:

  * Immunotoxins
  * Immunoconjugates
  * Antisense therapy
  * Peptide receptor antagonists
  * Interferons
  * Interleukins
  * Tumor-infiltrating lymphocytes
  * Lymphokine-activated killer cells
  * Gene therapy
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy

* No prior chemotherapy for GBM
* No other concurrent chemotherapy

Endocrine therapy

* Prior glucocorticoid therapy allowed
* No prior hormonal therapy for GBM
* Patients must be maintained on a stable corticosteroid regimen for at least 1 week

Radiotherapy

* No prior cranial irradiation
* No prior radiotherapy for GBM

Surgery

* Recovered from prior surgery

Other

* At least 1 week since prior treatment with any of the following:

  * Salicylates
  * Non-steroidal anti-inflammatory drugs
  * Sulfonamide medications
  * Vitamin C
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-07-12 (Actual); Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Response rate (complete and partial)

SECONDARY OUTCOMES:
Frequency of toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Jana Portnow, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (65):
- United States (65):
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Northwest Medical Specialist, PC, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Midwest Cancer Research Group, Incorporated, Skokie, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA at Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin